CLINICAL TRIAL: NCT03136861
Title: A 24-week, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Secukinumab in Controlling Spinal Pain in Patients With Axial Spondyloarthritis
Brief Title: SKIPPAIN - Speed of Onset of SecuKinumab-Induced Relief From Pain in Patients With AxIal SpoNdyloarthritis
Acronym: SKIPPAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457H3301; 2017-000401-21 (EudraCT Number)
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Spondyloarthritis
Keywords: axial spondyloarthritis; ankylosing spondylitis; non-radiographic axial spondyloarthritis; inflammatory back pain; spinal pain; secukinumab; AIN457
MeSH Terms: conditions — Spondylarthritis; Axial Spondyloarthritis; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Secukinumab 150 mg (Group A) (Experimental): Treatment Period 1: Secukinumab 150 mg (1 x 1.0 mL) s.c. administered at Baseline, Week 1, 2, 3 and 4
  Interventions: Biological: AIN457
- Placebo (Group B) (Placebo Comparator): Treatment Period 1: Placebo (1 x 1.0 mL) s.c. administered at Baseline and Week 1, 2, 3 and 4
  Interventions: Biological: AIN457; Drug: AIN457 Placebo
- Arm A1 (Active Comparator): Treatment Period 2: Secukinumab 150 mg (1 x 1.0 mL) plus placebo (1 x 1.0 mL) administered at Week 8, 12, 16 and 20
  Interventions: Biological: AIN457; Drug: AIN457 Placebo
- Arm A2 (Active Comparator): Treatment Period 2: Secukinumab 150 mg (1 x 1.0 mL) plus placebo (1 x 1.0 mL) administered at Week 8, 12, 16 and 20
  Interventions: Biological: AIN457; Drug: AIN457 Placebo
- Arm A3 (Active Comparator): Treatment Period 2: Secukinumab 300 mg (2 x 1.0 mL) administered at Week 8, 12, 16, and 20
  Interventions: Biological: AIN457
- Arm B1 (Active Comparator): Treatment Period 2: Secukinumab 150 mg (1 x 1.0 mL) plus placebo (1 x 1.0 mL) administered at Week 8, 12, 16 and 20
  Interventions: Biological: AIN457; Drug: AIN457 Placebo
- Arm B2 (Active Comparator): Treatment Period 2: Secukinumab 300 mg (2 x 1.0 mL) administered at Week 8, 12, 16, and 20
  Interventions: Biological: AIN457

INTERVENTIONS:
Biological: AIN457 — anti IL-17a monoclonal antibody
  Other Names: secukinumab
Drug: AIN457 Placebo — Placebo matching AIN457
  Other Names: Placebo
  Arms: Arm A1; Arm A2; Arm B1; Placebo (Group B)

SUMMARY:
The purpose of the study was to evaluate the efficacy and safety of secukinumab 150 mg compared to placebo in the early management (Baseline to Week 8) of spinal pain, disease activity, fatigue, and predictability of disease flares in patients with axial spondyloarthritis (axSpA) who had an inadequate response to prior non-steroidal anti-inflammatory drugs (NSAIDs). This study also explored the efficacy and safety of secukinumab 300 mg compared to secukinumab 150 mg from Week 8 to Week 24 in order to assess the potential additional benefits of dose escalation in patients with axSpA.

DETAILED DESCRIPTION:
The study consisted of 2 treatment periods: a double-blind, placebo-controlled period from Baseline to Week 8 (Treatment Period 1) and a double-blind secukinumab treatment period from Week 8 to Week 24 (Treatment Period 2).

At Baseline (Treatment Period 1), patients were randomized in a 3:1 ratio to either secukinumab 150 mg (Group A) or placebo (Group B). At Week 8 (Treatment Period 2), patients were re-randomized and re-assigned respectively to 1 of 5 treatment arms to receive either secukinumab 150 mg or secukinumab 300 mg.

Patients assigned to secukinumab 150 mg (Group A) at Baseline who were responders (i.e. spinal pain score < 4) at Week 8 continued on the same dose until Week 24 under 1 treatment arm (Arm A1). Patients assigned to secukinumab 150 mg at Baseline who were non-responders at Week 8 were re-randomized to 1 of 2 treatment arms: secukinumab 150 mg (Arm A2) or secukinumab 300 mg (Arm A3) from Week 8 to Week 24.

Similarly, patients assigned to placebo (Group B) at Baseline were re-randomized to 1 of 2 treatment arms: secukinumab 150 mg (Arm B1) or secukinumab 300 mg (Arm B2) from Week 8 until Week 24.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of axial spondylarthritis (axSpA, either ankylosing spondylitis or non radiographic axial spondylarthritis) according to ASAS axSpA classification criteria
* patients with back pain for at least 3 months and age of onset less than 45 years
* Active axSpA as assessed by total BASDAI score of at least 4 at Baseline.
* Spinal pain numeric rating scale score of more than 4 at Baseline.
* inadequate response to or failure to respond to at least 2 different NSAIDs at the highest recommended dose for at least 4 weeks in total prior to randomization

Key Exclusion Criteria:

* Chest X-ray or MRI with evidence of ongoing infectious or malignant process
* Patients previously treated with any biological immunomodulating agents, except those targeting tumor necrosis factor alpha.
* Patients who have been exposed to more than one anti-tumor necrosis factor alpha agent.
* Active ongoing inflammatory diseases other than axial spondyloarthritis
* Other ongoing mechanical diseases affecting the spine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Bulgaria (3):
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Croatia (3):
  - Novartis Investigative Site, Zagreb, HRV
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zagreb
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Plzen-Bory
  - Novartis Investigative Site, Prague
- Estonia (3):
  - Novartis Investigative Site, Pärnu
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (2):
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Kuovola
- Greece (4):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Dublin, Ireland
- Novartis Investigative Site, Verona, VR, Italy
- Latvia (2):
  - Novartis Investigative Site, Liepāja
  - Novartis Investigative Site, Riga
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Kaunas, LT
- Poland (6):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (4):
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
- Spain (12):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Elda, Alicante
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Galdakao, Bizkaia
  - Novartis Investigative Site, Torrelavega, Cantabria
  - Novartis Investigative Site, Plasencia, Extremadura
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Ourense, Galicia
  - Novartis Investigative Site, Torrejón de Ardoz, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
- Sweden (4):
  - Novartis Investigative Site, Stockholm, SE
  - Novartis Investigative Site, Danderyd
  - Novartis Investigative Site, Halmstad
  - Novartis Investigative Site, Härnösand
- Novartis Investigative Site, Basel, Switzerland
- United Kingdom (5):
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Warrington
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is commited to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
Time Frame: Upon request
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Poddubnyy D, Pournara E, Zielinska A, Baranauskaite A, Jimenez AM, Sadhu S, Schulz B, Rissler M, Perella C, Marzo-Ortega H. Rapid improvement in spinal pain in patients with axial spondyloarthritis treated with secukinumab: primary results from a randomized controlled phase-IIIb trial. Ther Adv Musculoskelet Dis. 2021 Oct 22;13:1759720X211051471. doi: 10.1177/1759720X211051471. eCollection 2021. PMID 34707696
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 66 centers in 17 countries worldwide: Spain(14), Czech Republic(3), Finland(2), Lithuania(2), Estonia(3), Latvia(3), Switzerland(1), Russia(4), Sweden(4), United Kingdom(5), Belgium(2), Ireland(2), Poland(7), Croatia(3), Bulgaria(5), Greece(5), Italy(1).
Pre-assignment Details: At Baseline, patients were randomized to either secukinumab 150 mg or placebo (Group A or B). At Week 8, patients were re-randomized or re-assigned respectively to 1 of 5 treatment arms to receive either secukinumab 150 mg or secukinumab 300 mg (Arm A1 to B2).
Period: Treatment Period 1 (TP1)(Baseline-Wk 8)
Arm/Group | Secukinumab 150 mg (Group A) | Placebo (Group B) | Arm A1 | Arm A2 | Arm A3 | Arm B1 | Arm B2
Started (All randomized patients were included in the Full Analysis Set (FAS) and Safety Analysis Set (SAF).) | 285 | 95 | 0 | 0 | 0 | 0 | 0
Completed | 278 | 89 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subject/Guardian Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Informed Consent | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (TP2) (Wk 8-Wk 24)
Arm/Group | Secukinumab 150 mg (Group A) | Placebo (Group B) | Arm A1 | Arm A2 | Arm A3 | Arm B1 | Arm B2
Started (All randomized patients were included in the Full Analysis Set (FAS) and Safety Analysis Set (SAF).) | 0 | 0 | 90 | 94 | 94 | 45 | 44
Completed | 0 | 0 | 88 | 93 | 92 | 45 | 43
Not Completed | 0 | 0 | 2 | 1 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Informed Consent | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: At Baseline Treatment Period 1, 380 patients were randomized to either secukinumab 150 mg or placebo (Group A or B). All the patients who completed Treatment Period 1 (367) were re-randomized or re-assigned respectively to 1 of 5 treatment arms to receive either secukinumab 150 mg or secukinumab 300 mg (Arm A1 to B2) in Treatment Period 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 150 mg (Group A) | Placebo (Group B) | Arm A1 | Arm A2 | Arm A3 | Arm B1 | Arm B2 | Total
Number analyzed (Participants) | 285 | 95 | 0 | 0 | 0 | 0 | 0 | 380
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age continuous at Baseline Treatment Period 1
  Years | 42.3 (11.88) | 40.9 (12.20) |  |  |  |  |  | 42.0 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at Baseline Treatment Period 1
  Participants
    Female | 106 | 39 |  |  |  |  |  | 145
    Male | 179 | 56 |  |  |  |  |  | 235
Race/Ethnicity, Customized [Number; unit: Participants] — Race at Baseline Treatment Period 1
  Participants
    Caucasian | 267 | 93 |  |  |  |  |  | 360
    Asian | 2 | 1 |  |  |  |  |  | 3
    Other | 16 | 1 |  |  |  |  |  | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Spinal Pain Numerical Rating Scale (NRS) Score Below 4 at Week 8 (Treatment Period 1)
Description: The spinal pain numerical rating scale (NRS) is an 11-point scale to assess pain intensity in patients who are able to self-report. It is an 11-point scale from 0-10: 1) "0" = no pain. 2) "10" = the most intense pain imaginable. To calculate the average spinal pain, the patient was asked to answer 2 questions to get 2 pain ratings, the total spinal pain corresponding to the intensity of spinal pain experienced on an average over 24 hours during the previous week and the nocturnal back pain corresponding to the intensity of spinal pain experienced on an average over the night during the previous week.
Time Frame: Week 8
Population: Full Analysis Set (FAS) in Treatment Period 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg (Group A) | Placebo (Group B)
Number analyzed (Participants) | 279 | 92
Participants
  Average Spinal Pain Score: Yes | 91 | 19
  Average Spinal Pain Score: No | 188 | 73
  Total Spinal Pain Score: Yes | 77 | 17
  Total Spinal Pain Score: No | 202 | 75
  Nocturnal Spinal Pain Score: Yes | 92 | 16
  Nocturnal Spinal Pain Score: No | 187 | 76
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group A) vs Placebo (Group B); Average Spinal Pain Score <4 at Week 8; Test type: Superiority; p = 0.0264, Regression, Logistic; Logistic regression model: logit (proportion) = treatment + stratification factor of prior exposure to TNF inhibitors (i.e. TNF-naïve or TNFα-IR); Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.08 to 3.33]
Statistical Analysis 2: Comparison: Secukinumab 150 mg (Group A) vs Placebo (Group B); Total Spinal Pain Score <4 at Week 8; Test type: Superiority; p = 0.0720, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.95 to 3.10]
Statistical Analysis 3: Comparison: Secukinumab 150 mg (Group A) vs Placebo (Group B); Nocturnal Spinal Pain Score; Test type: Superiority; p = 0.0043, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.38, 95% CI 2-sided [1.31 to 4.31]

2. Secondary Outcome: Percentage of Participants With a Bath Ankylosing Spondylitis Disease Activity Index Score Below 4 at Week 8 (Treatment Period 1)
Description: The Bath ankylosing spondylitis disease activity index (BASDAI) consists of a 0 through 10 scale, which is used to answer 6 questions pertaining to the 5 major symptoms of ankylosing spondylitis. To give each symptom equal weighting, the mean (average) of the 2 scores relating to morning stiffness (questions 5 and 6) is taken. The mean of questions 5 and 6 is added to the scores from questions 1-4. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score.
Time Frame: Week 8
Population: Full Analysis Set (FAS) in Treatment Period 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg (Group A) | Placebo (Group B)
Number analyzed (Participants) | 280 | 92
Participants
  Yes (n=95,22) | 95 | 22
  No (n=185,70) | 185 | 70
Statistical Analysis 1: Comparison: Secukinumab 150 mg (Group A) vs Placebo (Group B); BASDAI Score <4 at Week 8; Test type: Superiority; p = 0.0466, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.01 to 3.04]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from first dose of study treatment until end of study treatment plus 12 weeks, up to a maximum duration of 32 weeks.
Description: Any sign or symptom that occurs after written informed consent provided. Treatment emergent adverse events were reported until end of study treatment plus 12 weeks post treatment.
  Treatment emergent adverse events occurring during Treatment Period 1 are recorded in Group A and B arms.
  Treatment emergent adverse events occurring during Treatment Period 2 are recorded in Arm A1 to Arm B2.
Arm/Group | Secukinumab 150 mg (Group A) | Placebo (Group B) | Arm A1 | Arm A2 | Arm A3 | Arm B1 | Arm B2
All-Cause Mortality (participants affected / at risk) | 0/285 | 0/95 | 0/90 | 0/94 | 0/94 | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 4/285 | 0/95 | 3/90 | 1/94 | 1/94 | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 59/285 | 23/95 | 21/90 | 24/94 | 23/94 | 9/45 | 13/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg (Group A) (N=285) | Placebo (Group B) (N=95) | Arm A1 (N=90) | Arm A2 (N=94) | Arm A3 (N=94) | Arm B1 (N=45) | Arm B2 (N=44)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg (Group A) (N=285) | Placebo (Group B) (N=95) | Arm A1 (N=90) | Arm A2 (N=94) | Arm A3 (N=94) | Arm B1 (N=45) | Arm B2 (N=44)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 0 | 0 | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Fatigue (General disorders) | 6 | 0 | 1 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 0 | 0 | 0 | 3 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | 2 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 1 | 1 | 3 | 4 | 2 | 2
Otitis externa (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 3 | 0 | 2 | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 1 | 0 | 3 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 2 | 1 | 0
Blood creatinine increased (Investigations) | 4 | 0 | 3 | 1 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 3 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 10 | 1 | 2 | 2 | 3 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 3 | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 1 | 0 | 2 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 4 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03136861/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT03136861/SAP_000.pdf